CLINICAL TRIAL: NCT06700330
Title: Study of the Etiology, Clinical Picture, Complications and Outcomes of Necrotizing Pancreatitis in Children.
Brief Title: Etiology, Clinical Picture, Complications and Outcomes of Necrotizing Pancreatitis in Children.
Status: Completed | Type: Observational
Sponsor: Moscow Regional Research and Clinical Institute (MONIKI) (Other Government)
Responsible Party: Sponsor
Other Study IDs: 16/01.11.2024
Record Dates: First submitted 2024-11-20; First posted 2024-11-21 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Pancreatitis; Pancreatitis, Acute Necrotizing; Children
Keywords: Pancreatitis; Acute Necrotizing Pancreatitis; Children
MeSH Terms: conditions — Pancreatitis; Pancreatitis, Acute Necrotizing | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Children with necrotizing pancreatitis: children who have suffered acute pacreatitis
  Interventions: Other: no intervention, observational study

INTERVENTIONS:
Other: no intervention, observational study — Only data from the patient file.

SUMMARY:
The aim of this research is to study the etiology, the clinical picture, the management, the complications and the outcomes of necrotic pancreatitis in children.

Currently, there is a significant number of errors in the early diagnosis of AP in children associated with the complexity of differential diagnosis, which leads to the untimely verification of the correct diagnosis and, consequently, to incorrect treatment tactics, which could be accompanied by an increase in the severe forms of the disease and an increase in mortality.

DETAILED DESCRIPTION:
Acute pancreatitis (AP) is an acute inflammatory disease of the exocrine pancreas. Clinical manifestations vary from mild abdominal discomfort to metabolic disorders, sepsis, fluid sequestration, multiple organ failure and death. According to the international data, the annual incidence of AP in children is 3-13 cases per 100,000 people, but in recent years, there has been an increase in the incidence of this pathology. Necrotic pancreatitis in children accounts for up to 25-30% of the cases of all forms of AP. Despite the successes achieved in the diagnosis and treatment of AP, the mortality rate for this pathology is up to 5%, according to various authors. In addition, given the varying degrees of the prevalence of the destructive process in the pancreas and the parapancreatic tissue, the choice of surgical treatment still remains a subject of discussion. The treatment of moderately severe (MSAP) and severe (SAP) necrotic pancreatitis is a complex task due to the variety of causes of the disease, the incompletely understood pathogenesis and the uncertainty in predicting the results.

Paralytic ileus with the development of intestinal failure is the main pathogenetic factor in the development of a septic condition in AP, but there is tendency of insufficient attention being paid to this fact in pediatric practice, which determines the lack of a unified approach to the treatment of intestinal failure syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Consent of the patient or legal representative
* Age from 0-18 years
* Moderate severe (MSAP) or severe acute pancreatitis (SAP) according to Atlanta criteria revisited in 2012
* Acute Pancreatitis was established in the presence of at least two of three criteria according to the classification developed by the INSPPIRE group (International Study Group of Pediatric Pancreatitis: In Search for a Cure): abdominal pain corresponding to the diagnostic hypothesis; an increase in amylase and / or lipase in the blood serum by ≥3 times; imaging findings characteristic of AP: abdominal ultrasound and/or contrast-enhanced CT.

Exclusion Criteria:

* mild acute pancreatitis
* chronic pancreatitis
* no consent from patient or legal representative

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Moscow Regional Scientific Research Clinical Institute named after M.F. Vladimirsky
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-02-18 (Actual)

PRIMARY OUTCOMES:
the frequency of occurrence of various etiologic causes of necrotizing pancreatitis in children | From enrollment to the end of treatment (2 month)
  based on the study, the most common causes of necrotizing pancreatitis in children will be identified

SECONDARY OUTCOMES:
The duration from the onset of the disease to the start of the treatment | from the onset of the disease to the end of treatment (up to 20 weeks)
The duration of hospital stay | from admission to hospital until the end of treatment (up to 8 weeks)
  the effect of each risk factor on the duration of hospital stay
The length of ICU stay | During ICU stay (up to 60 days)
The effect of comorbidities on the severity of the disease | from admission to hospital until the end of treatment (up to 8 weeks)
Intestinal failure | from admission to hospital until the end of treatment (up to 8 weeks)
  the effect of Intestinal failure on the duration of hospital stay
Paralytic ileus | from admission to hospital until the end of treatment (up to 8 weeks)
  the effect of paralytic ileus on the severity of acute pancreatitis and the length of hospital stay
Mortality | from admission to hospital until the end of treatment (up to 20 weeks)
Enzymatic parapancreatitis | from admission to hospital until the end of treatment (up to 10 weeks)
  the effect on severity of the disease and the outcome
Purulent-necrotic parapancreatitis | from admission to hospital until the end of treatment (up to 20 weeks)
  the effect on severity of the disease and the outcome
Biliary obstruction | from admission to hospital until the end of treatment (up to 20 weeks)
Surgical interventions | from admission to hospital until the end of treatment (up to 20 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Dmitriy A Pyhteev, PhD, Study Director — Head of the Department of Pediatric Surgery; Leonid M Elin, Principal Investigator — Moscow Regional Scientific Research Clinical Institute named after M.F. Vladimirsky
Locations (1):
- Moscow Regional Scientific Research Clinical Institute named after M.F. Vladimirsky, Moscow, Moscow Oblast, Russia

IPD SHARING:
Plan to Share IPD: Yes
A complete dataset can be provided upon reasoned request